CLINICAL TRIAL: NCT05871437
Title: Prospective, Multicenter, Randomized Controlled Clinical Trial on the Effect of Huaier Granules in Reducing Tumor Marker Levels in Patients With Early-Stage Breast Cancer
Brief Title: Randomized Controlled Clinical Study on the Reduction of Tumor Marker Levels in Breast Cancer Patients by Huaier Granules
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Fudan University (Other)
Collaborators: LinkDoc Technology (Beijing) Co. Ltd. (Industry); Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Zhimin Shao, professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HE- 202504
Record Dates: First submitted 2023-05-04; First posted 2023-05-23 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
Keywords: Huaier granule; breast cancer; level of tumor markers
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Huaier Granule+Conventional clinical therapeutic drugs (Experimental): Huai er Granules: Oral administration, 10g each time, three times a day, for one year. In case of intolerable toxicity, withdrawal from the study for any reason, or death, the first occurrence shall prevail. Or the researchers determine that they will no longer benefit. For specific usage, please refer to the drug instructions. For specific usage, please refer to the drug instructions.
  Interventions: Drug: Huaier granule
- Conventional clinical therapeutic drugs (No Intervention): Treatment and follow-up were carried out in accordance with clinical routines

INTERVENTIONS:
Drug: Huaier granule — On the basis of routine clinical treatment/follow-up, take Huaier Granules orally, 10g each time, three times a day, for one year continuously or until disease progression, intolerable toxicity, withdrawal from the study for any reason or death occurs, whichever occurs first.
  Other Names: Z20000109（NMPA Approval Number）
  Arms: Huaier Granule+Conventional clinical therapeutic drugs

SUMMARY:
This study is a prospective, multicenter, randomized controlled clinical trial designed to evaluate the rate of reduction of tumor markers to normal levels in breast cancer patients treated with Huaier granules compared to the control group.

DETAILED DESCRIPTION:
This study is a prospective, multicenter, randomized controlled clinical trial. Patients in the follow-up phase after breast cancer surgery were screened, excluding those with recurrence or metastasis, while having tumor markers (CEA/CA125/CA153) levels exceeding the upper limit of normal. A total of 232 patients were enrolled and randomly assigned to either the control group or the experimental group. They were followed up for one year, or until intolerable toxicity, withdrawal from the study for any reason, or death, whichever occurred first; or until the investigator determined that no further benefit could be obtained.

During the entire study period, the planned patient recruitment and enrollment duration is approximately 12 months, with a total follow-up duration of 12 months per participant. After enrollment, patients will be followed up every three months until the study concludes, or until the patient withdraws from the study for any reason or passes away.

ELIGIBILITY:
Inclusion Criteria:

* 18 ≤ age ≤ 75 years old, regardless of gender.
* Postoperative pathological diagnosis of breast cancer.
* Imaging or pathological examination without evidence of recurrence or metastasis.
* If tumor markers are elevated, it is necessary to go to the corresponding department for medical treatment or issue a corresponding examination when necessary to exclude recurrence, metastasis or the second primary tumor of breast cancer.
* One or more tumor markers in CEA/CA125/CA153 exceed the upper limit of normal values.
* The liver and kidney functions meet the following conditions: AST and ALT< 3 ULN, total bilirubin ≤ 2 ULN, and blood creatinine<1.5 ULN;
* Other laboratory tests meet the following requirements: Hb ≥ 9g/dl, platelet count ≥ 60 × 10^9/L, absolute neutrophil count>1.0 × 10^9/L.
* The patient's ECOG physical state score is 0 or 1.
* The subjects participated in this study voluntarily and signed an informed consent form.

Exclusion Criteria:

* Diagnosed as any other malignant tumor within the 5 years prior to enrollment, except for malignant tumors with low risk of metastasis and death (5-year survival rate>90%), such as fully treated basal cell or squamous cell skin cancer or cervical cancer in situ.
* Imaging or pathological confirmation of recurrence and metastasis.
* Serious infections (CTCAE>Level 2) occurred within the first 4 weeks of enrollment, such as severe pneumonia, bacteremia, and infection complications that require hospitalization; Symptoms and signs of infection or the need for oral or intravenous antibiotic treatment within 2 weeks prior to enrollment, excluding the use of prophylactic antibiotics.
* Suffering from severe acute and chronic diseases.
* Suffering from severe diabetes whose blood sugar cannot be effectively controlled.
* Patients who are unable to take oral medication, those who are allergic to the ingredients of Huaier granules, and pregnant or lactating women.
* Drug abusers, or those who suffer from psychological or mental illnesses that may interfere with research compliance.
* The researcher believes that it is not suitable to participate in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Recovery rate of any tumor marker (CEA/CA125/CA153) to normal | Start of treatment until 2-year follow-up
  The rate at which one or more tumor markers (CEA/CA125/CA153) exceed the upper limit of normal values before patient enrollment and any tumor marker that rises before enrollment decreases to the normal range after the end of Huaier Granule treatment

SECONDARY OUTCOMES:
The incidence and severity of adverse events (AE) and severe adverse events (SAE) | Start of treatment until 2-year follow-up
  The definition and severity grading of AE and SAE refer to the corresponding descriptions in the definition and evaluation section of adverse events, and the incidence rate is defined as the proportion of patients with AE and SAE to the corresponding total population
The incidence and severity of adverse reaction (ADR), severe adverse reactions(SADR), suspicious and unexpected severe adverse reaction (SUSAR) | Start of treatment until 2-year follow-up
  The definition and severity grading of ADR, severe ADR, and SUSAR refer to the corresponding descriptions in the definition and evaluation section of adverse events. The incidence rate is defined as the proportion of patients with ADR, severe ADR, and SUSAR to the corresponding total population
Quality of Life Score | Start of treatment until 2-year follow-up
  Evaluation using the EORTC QLQ-C30 (Chinese version) core quality of life scale developed by the European Organization for Cancer Research and Treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Zhimin Shao, PhD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No